CLINICAL TRIAL: NCT01650389
Title: Phase II Randomised Controlled Trial to Evaluate Safety and Immunogenicity of MVA85A and Selective, Delayed Bacille Calmette-Guerin (BCG) Vaccination in Infants of HIV Infected Mothers
Brief Title: Safety and Immunogenicity of MVA85A Prime and Bacille Calmette-Guerin Boost Vaccination
Acronym: MVA(TB)029
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mark Hatherill (Other)
Collaborators: Medical Research Council (Other Government); Wellcome Trust (Other); Department for International Development, United Kingdom (Other Government); University of Oxford (Other); University of Stellenbosch (Other); Oxford-Emergent Tuberculosis Consortium (Unknown)
Responsible Party: Sponsor-Investigator, Mark Hatherill, Associate Professor, University of Cape Town
Organization: University of Cape Town (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: G1100570/1; G1100570 (Other Grant/Funding Number: Medical Research Council (UK))
Record Dates: First submitted 2012-07-23; First posted 2012-07-26 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Tuberculosis; HIV
Keywords: Tuberculosis; HIV; BCG; Infant
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MVA85A (Experimental): 1 x 10(superscript'8') pfu MVA85A vaccine intradermal within 96 hours of birth
  Interventions: Biological: MVA85A; Biological: BCG Vaccine SSI
- Candin (Active Comparator): Equal volume intradermal administration within 96 hours of birth
  Interventions: Biological: Candin; Biological: BCG Vaccine SSI

INTERVENTIONS:
Biological: MVA85A
  Arms: MVA85A
Biological: Candin
  Arms: Candin
Biological: BCG Vaccine SSI — All infants who test negative by HIV PCR will receive BCG vaccination at 8 weeks of age.
  Infants who test positive by HIV PCR will not receive BCG vaccination.

SUMMARY:
Rationale: The Bacille Calmette-Guérin (BCG) vaccine protects children against disseminated tuberculosis (TB) including TB meningitis and miliary TB, but efficacy against pulmonary TB is inconsistent among children and adults. Administration of live attenuated BCG to infants known to be HIV infected is contraindicated by the World Health Organization (WHO), due to the risk of serious vaccine adverse events (BCG disease. Developing countries, which lack capacity for integration of early infant HIV testing with infant vaccination schedules, have not fully implemented the WHO guidelines on BCG vaccination of HIV exposed infants. Newborn infants of HIV infected mothers continue to receive routine BCG before HIV infection has been excluded.

Clinical trials of new viral-vectored TB vaccines, including MVA85A, a modified vaccinia virus Ankara (MVA) vaccine expressing the Mycobacterium tuberculosis antigen 85A, have to date enrolled infants who were already vaccinated with routine BCG at birth. However, TB vaccination regimens that depend on newborn BCG will remain unsafe for HIV infected infants. Infants of HIV infected mothers, who constituted 29% of babies born in South Africa in 2009, would benefit from a new TB vaccination strategy, in which BCG is delayed until after HIV infection has been excluded. These HIV exposed infants also have greater increased risk of TB disease. Testing the safety and immunogenicity of MVA85A vaccine prime, followed by selective delayed BCG boost, in HIV exposed newborns, is a critical step towards delivery of a new TB vaccine regimen that is safe and effective for all infants, regardless of HIV exposure.

Study Design: Double blinded, randomised, controlled trial. HIV exposed infants will be randomised 1:1 to receive single dose, intradermal MVA85A vaccine or Candin® control at birth. The first 60 infants enrolled in the trial will form a pilot safety cohort for formal Data Monitoring & Ethics Committee (DMEC) safety review. Thereafter, safety and immunogenicity outcomes will be measured in all infants.

Study Population: Infants (n=340) born to HIV infected mothers receiving antiretroviral therapy (ART) or Prevention of Mother to Child Transmission (PMTCT) prophylaxis.

Sites: Worcester (University of Cape Town) and Khayelitsha (Stellenbosch University), South Africa

Study Intervention: Newborn infants will receive 1 x 108 pfu MVA85A vaccine or Candin® control by intradermal injection. Infants confirmed HIV uninfected by HIV PCR will receive BCG Vaccine SSI at 8 weeks of age. Infants confirmed HIV infected by HIV PCR will not receive BCG.

Primary specific aims:

To evaluate the safety of MVA85A given at birth to HIV exposed uninfected infants.

To evaluate the safety of BCG given at 8 weeks of age to HIV exposed uninfected infants, using an MVA85A prime and BCG boost strategy.

Secondary specific aims:

To evaluate the immunogenicity of MVA85A given at birth to HIV exposed uninfected infants.

To evaluate the immunogenicity of BCG given at 8 weeks of age to HIV exposed uninfected infants, using an MVA85A prime and BCG boost strategy.

Safety endpoints:

Local, regional, and systemic adverse events (AEs) and serious adverse events (SAEs).

Immunology endpoints:

Frequencies of CD4 and CD8 T cells producing any of 4 cytokines (IL-17, IFN-γ, TNF-α, or IL-2), or polyfunctional combinations of these cytokines simultaneously, following stimulation with antigen Ag85A or BCG, measured by whole blood intracellular cytokine assay (WB-ICS).

Specific proliferative capacity of CD8 and CD4 T cells that produce any of the three cytokines (IFN-γ, TNF-α, and/or IL-2) or combinations of these cytokines simultaneously, measured by a novel whole blood 6-day lymphoproliferative flow cytometric assay (WB-prolif).

Relative proportions and absolute numbers of peripheral blood myeloid and lymphoid cell subsets, measured directly ex vivo by flow cytometry.

Study groups: The first 60 infants enrolled in Study Group 1 will undergo intensive safety evaluation, followed by DMEC review of Day-28 safety data. The DMEC will make a formal recommendation on continuation of enrollment and/or changes to the protocol, based on this safety review. Study Groups 2-5 will be evaluated for clinical safety and immunology outcomes.

Statistical Analysis: Cumulative 12-month incidence of local, regional, and systemic AEs, by category, will be compared for HIV exposed uninfected subjects receiving MVA85A vaccine or Candin® control at birth. The sample size has 90% probability of detecting an SAE with a true occurrence rate of 1.5% in infants receiving MVA85A vaccine and 80% power to detect a 15% difference in the rate of non-serious AEs (20% compared to 35%) between the two study arms (p<0.05). Multivariate models will be built to explore longitudinal immunological data and identify independent associations with MVA85A vaccination and covariates of interest.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected mother receiving either cART, or started on PMTCT prophylaxis
* Maternal antenatal and post-natal written informed consent;
* Maternal age 18 years or older at the time of informed consent;
* Infant age < 96 hours;
* Infant birth and residence in the study area;
* Mother contactable and able to attend follow-up visits.

Exclusion Criteria:

* Neonatal Apgar score < 7 at 5 minutes;
* Infant birth weight < 2,000g or > 4,500g;
* Estimated infant gestational age < 32 weeks;
* Neonatal respiratory distress;
* History or evidence of infant congenital abnormality, or immunosuppressive condition, other than HIV infection;
* Any maternal or infant condition or systemic illness that in the opinion of the investigator is likely to affect safety or immunogenicity of study vaccine;
* Infant BCG vaccination prior to enrollment;
* Residence in a household, or frequent close contact, with an adult diagnosed with active TB who has not yet completed TB treatment;
* Mother with active TB who has not yet completed TB treatment;
* Unknown or negative maternal HIV status;
* Intention to leave the study area and/or unable to attend follow-up visits.

Max Age: 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 248 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Safety | 1 year
  Local, regional, and systemic adverse events (AEs) and serious adverse events (SAEs).

SECONDARY OUTCOMES:
Immunogenicity | 1 Year
  Frequencies of CD4 and CD8 T cells producing IL-17, IFN-γ, TNF-α, or IL-2, or polyfunctional combinations of these cytokines, following stimulation with antigen Ag85A or BCG, measured by whole blood intracellular cytokine assay.
  Specific proliferative capacity of CD8 and CD4 T cells that produce IFN-γ, TNF-α, or IL-2, or combinations of these cytokines, measured by whole blood 6-day lymphoproliferative flow cytometric assay.
  Relative proportions and absolute numbers of peripheral blood myeloid and lymphoid cell subsets, measured directly ex vivo by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hatherill, MD, FCPaed, Principal Investigator — University of Cape Town
Locations (2):
- South Africa (2):
  - Desmond Tutu TB Centre (DTTC), Stellenbosch University, Khayelitsha
  - South African Tuberculosis Vaccine Initiative (SATVI), University of Cape Town, Worcester

REFERENCES:
- [Derived] Nemes E, Hesseling AC, Tameris M, Mauff K, Downing K, Mulenga H, Rose P, van der Zalm M, Mbaba S, Van As D, Hanekom WA, Walzl G, Scriba TJ, McShane H, Hatherill M; MVA029 Study Team. Safety and Immunogenicity of Newborn MVA85A Vaccination and Selective, Delayed Bacille Calmette-Guerin for Infants of Human Immunodeficiency Virus-Infected Mothers: A Phase 2 Randomized, Controlled Trial. Clin Infect Dis. 2018 Feb 1;66(4):554-563. doi: 10.1093/cid/cix834. PMID 29028973